CLINICAL TRIAL: NCT01907828
Title: A Feasibility Study to Evaluate the Effect of Concomitant Renal Denervation and Cardiac Ablation on AF Recurrence
Acronym: RDN+AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJM-CIP-0009
Record Dates: First submitted 2013-07-17; First posted 2013-07-25 (Estimated); Results first posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Persistent Atrial Fibrillation; Paroxysmal Atrial Fibrillation; Hypertension
MeSH Terms: conditions — Atrial Fibrillation; Hypertension | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cardiac ablation + renal artery ablation (Experimental): Renal artery ablation with the EnligHTN™ Renal Denervation System
  Interventions: Device: Renal Artery Ablation; Device: Cardiac Ablation
- Cardiac ablation (Active Comparator): Cardiac ablation
  Interventions: Device: Cardiac Ablation

INTERVENTIONS:
Device: Renal Artery Ablation — Renal artery denervation using the EnligHTN™ Renal Denervation System
  Arms: Cardiac ablation + renal artery ablation
Device: Cardiac Ablation — Safire BLU™ Duo or Therapy Cool Path Duo Irrigated Ablation Catheter or Therapy Cool Flex Irrigated Ablation Catheter EnSite Velocity System Agilis NxT Guiding Introducer

SUMMARY:
The purpose of this post market clinical investigation is to complete preliminary evaluation on whether or not concomitant renal denervation with the EnligHTN™ Renal Denervation System and cardiac ablation will result in improved outcomes as compared to ablation alone in patients with uncontrolled hypertension being treated for Atrial Fibrillation

DETAILED DESCRIPTION:
This is a post market, prospective, multicenter, 2:1 randomized study of the EnligHTN™ Renal Denervation System in conjunction with atrial fibrillation ablation. Up to one hundred subjects with paroxysmal or persistent atrial fibrillation and uncontrolled hypertension will be enrolled in the study. All subjects will undergo cardiac ablation for the treatment of atrial fibrillation. Per the 2:1 randomization, a minimum of 50 or 2/3 of the total patient cohort will also undergo renal artery ablation. Subjects will be followed up to years (2) years post procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age at time of consent
* Subject must be able and willing to provide written informed consent
* Subject must be able and willing to comply with the required follow-up schedule
* Subject is a candidate for catheter ablation for the treatment of paroxysmal or persistent atrial fibrillation as per the hospital standard of care
* Subject has office Systolic Blood Pressure ≥ 140 mmHg at baseline visit
* Subject has a daytime mean Systolic Ambulatory Blood Pressure > 135 mmHg within 90 days prior to procedure
* Subject has established hypertension (diagnosed ≥12 month prior to baseline) and is taking >3 anti-hypertensive medications, including 1 diuretic
* Subject has been on a stable unchanged anti-hypertensive medication regimen for a minimum of 4 weeks prior to the ablation procedure

Exclusion Criteria:

* Subject has long standing atrial fibrillation
* Subject has had a previous ablation for atrial fibrillation
* Subject has had a previous renal denervation procedure
* Subject has had a CABG procedure within the last 180 days (six months)
* Subject has a left atrial thrombus
* Subject has a contraindication to anticoagulation (i.e. heparin or warfarin)
* Subject has unstable angina
* Subject has had a myocardial infarction within the previous two months
* Subject has a left ventricular ejection fraction (LVEF) <40% as determined by pre-procedure TTE
* Subject has significant renovascular abnormalities such as renal artery stenosis > 30%
* Subject has undergone prior renal angioplasty, renal denervation, indwelling renal stents, and/or abdominal aortic stent grafts
* Subject has hemodynamically significant valvular heart disease as determined by study investigator
* Subject has a life expectancy less than 12 months, as determined by the study investigator
* Subject is participating in another clinical study which has the potential to impact his/her hypertension or atrial fibrillation management (pharmaceutical/device/homeopathic)
* Subject is pregnant, nursing, or of childbearing potential and is not using adequate contraceptive methods
* Subject has active systemic infection
* Subject has renal arteries < 4 mm in diameter
* Subject has an estimated GFR <45 mL/min per 1.73 m2 using the Modification of Diet in Renal Disease (MDRD) formula
* Subject had a renal transplant or is awaiting a renal transplant
* Subject has blood clotting or bleeding abnormalities
* Subject has secondary arterial hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-04-15 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Piorkowski, MD, Principal Investigator — Herzzentrum Dresden GmbH Universitätsklinik
Locations (2):
- Germany (2):
  - Herzzentrum Dresden GmbH Universitätsklinik, Dresden
  - Herzzentrum Leipzig GmbH, Leipzig

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kirstein B, Tomala J, Mayer J, Ulbrich S, Wagner M, Pu L, Piorkowski J, Hankel A, Huo Y, Gaspar T, Richter U, Hindricks G, Piorkowski C. Effect of concomitant Renal DeNervation and cardiac ablation on Atrial Fibrillation recurrence - RDN+AF study. J Cardiovasc Electrophysiol. 2023 Jan;34(1):44-53. doi: 10.1111/jce.15714. Epub 2022 Dec 1. PMID 36259713

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrollment was completed with a total of 61 participants randomized at 2 sites in Germany. The first and last participants were enrolled on May 12, 2014, and July 21, 2016, respectively.
Groups:
- Renal Artery Ablation + Cardiac Ablation (RDN+AF): Participants treated with renal artery ablation using the EnligHTN System and cardiac ablation.
- Cardiac Ablation (AF): Participants treated with cardiac ablation alone.
Period: Overall Study
Arm/Group | Renal Artery Ablation + Cardiac Ablation (RDN+AF) | Cardiac Ablation (AF)
Started | 39 | 22
Underwent Procedure | 39 | 20 (2 participants terminated early)
1-month Follow-up | 37 (2 participants terminated early) | 17 (3 participants terminated early)
3-month Follow-up | 36 (1 participant terminated early) | 16 (1 participant terminated early)
6-month Follow-up | 35 (1 participant terminated early) | 16
12-month Follow-up | 34 (1 participant terminated early) | 16
24-month Follow-up | 32 (2 participants terminated early) | 16
Completed | 32 | 16
Not Completed | 7 | 6
Not completed — Exclusion criteria not met | 0 | 1
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Lost to Follow-up | 3 | 0
Not completed — Participant refused 24-month follow-up | 1 | 0
Not completed — Participant met exclusion criteria | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Renal Artery Ablation + Cardiac Ablation (RDN+AF) | Cardiac Ablation (AF) | Total
Number analyzed (Participants) | 39 | 22 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (7.9) | 63.0 (9.9) | 65.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 10 | 29
  Male | 20 | 12 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 39 | 22 | 61
Height [Mean (Standard Deviation); unit: cm] | 172.7 (10.1) | 173.6 (9.4) | 173.0 (9.8)
Weight [Mean (Standard Deviation); unit: kg] | 95.4 (17.9) | 93.7 (19.1) | 94.8 (18.2)
Body mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.9 (5.0) | 31.0 (5.4) | 31.6 (5.1)
Office Blood Pressure [Mean (Standard Deviation); unit: mmHg]
  Office Systolic Blood Pressure | 162.0 (18.6) | 167.1 (18.5) | 163.9 (18.5)
  Office Diastolic Blood Pressure | 87.5 (14.1) | 91.4 (10.6) | 88.9 (13.0)
Office Heart Rate [Mean (Standard Deviation); unit: beats per minute (bpm)] | 81.3 (23.9) | 76.7 (19.5) | 79.7 (22.4)
Number of Participants with a history of renal assessment prior to enrollment [Count of Participants; unit: Participants] — Renal artery imaging was performed using Computed Tomography (CT) or Magnetic Resonance (MR) angiogram within 90 days prior to enrollment. Non-contrast Magnetic Resonance Imaging (MRI) and doppler evaluation or ultrasound were also acceptable.
  Renal artery evaluation data collected included but was not limited to:
  * Type of evaluation (CT, MR angiogram, non-contrast MRI, doppler)
  * Length of artery(s)
  * Diameter of artery(s)
  * Number of main renal arteries
  * Number of accessory renal arteries
  * Presence and percent of stenosis
  * Other abnormalities
  Participants | 2 | 0 | 2
New York Heart Association (NYHA) Class of Cardiac Disease [Count of Participants; unit: Participants] — NYHA assessment was evaluated based on limitation of physical activity using the following definitions:
  Class I - Patients with cardiac disease but resulting in no limitation of physical activity.
  Class II- Patients with cardiac disease resulting in slight limitation of physical activity.
  Class III - Patients with cardiac disease resulting in marked limitation of physical activity.
  Class IV- Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort.
  Class I was considered to have better outcomes and Class IV with worse outcomes.
  Participants
    Class I | 10 | 11 | 21
    Class II | 24 | 10 | 34
    Class III | 5 | 1 | 6
    Class IV | 0 | 0 | 0
Medical History [Count of Participants; unit: Participants]
  Myocardial Infarction | 1 | 3 | 4
  Coronary Artery Disease | 5 | 7 | 12
  Valvular Disease | 27 | 15 | 42
  Arrhythmia | 39 | 22 | 61
  Cardiomyopathy | 2 | 1 | 3
  Neurological events/Dysfunction | 2 | 2 | 4
  Hyperlipidemia | 20 | 11 | 31
  Diabetes | 16 | 7 | 23
  Smokers | 17 | 4 | 21
  Significant Alcohol Intake | 6 | 0 | 6
  Obstructive Sleep Apnea | 3 | 1 | 4
  Thyroid Disease | 8 | 6 | 14
  Liver Disease | 2 | 4 | 6
  Other Additional Medical History | 38 | 18 | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Freedom From Atrial Fibrillation at 12 Month
Description: The freedom from atrial fibrillation was assessed based on electrocardiographic data during nine months following the blanking period including the one week recording coinciding with the 12 month follow-up visit (9 months following the 3 month blanking period).
Time Frame: 12 months
Population: Data not collected from all participants: data were available for only 28 participants in the RDN+AF group, and 12 participants in the AF group
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Artery Ablation + Cardiac Ablation (RDN+AF) | Cardiac Ablation (AF)
Number analyzed (Participants) | 28 | 12
Participants | 16 | 4
Statistical Analysis 1: Comparison: Renal Artery Ablation + Cardiac Ablation (RDN+AF) vs Cardiac Ablation (AF); Kaplan-Meier analysis performed to provide freedom from atrial fibrillation rates at one year for each randomization arm using date of ablation procedure to date of first event; Test type: Other; p = 0.22, Log Rank

2. Secondary Outcome: Major Adverse Cardiac Events (MACE)
Description: Major adverse cardiac events (MACE) were summarized as a percentage based on number of subjects at baseline for each group (RDN+AF group = 39, AF group = 22).
Time Frame: 7 days, 6 months, 12 months, and 24 months post procedure
Population: For each group, the outcome measure was analyzed in participants randomized at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Artery Ablation + Cardiac Ablation (RDN+AF) | Cardiac Ablation (AF)
Number analyzed (Participants) | 39 | 22
Participants
  MACE within 7 days of procedure | 0 | 2
  MACE within 6 months of procedure | 0 | 2
  MACE within 12 months of procedure | 0 | 2
  MACE within 24 months of procedure | 0 | 2

3. Secondary Outcome: Percentage of Participants Who Experience Peri-procedural Events
Description: Peri-procedural events within 30 days post procedure were summarized as a percentage based on the number of subjects at baseline for each group (RDN+AF group= 39, AF group=22)
Time Frame: 30 days post procedure
Population: Peri-procedural events within 30 days post procedure were summarized as a percentage based on the number of subjects at baseline for each group (RDN+AF group= 39, AF group=22).
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Artery Ablation + Cardiac Ablation (RDN+AF) | Cardiac Ablation (AF)
Number analyzed (Participants) | 39 | 22
Participants
  Cardiac Arrest | 0 | 1
  Pericardial Effusion | 0 | 1
  Paroxysmal Atrial Tachycardia | 1 | 0
  Hematoma | 0 | 1
  Pericardial Tamponade | 0 | 1
  Bleeding | 0 | 1
  VASC Pseudoaneurysm | 1 | 0
  Air Embolus | 3 | 0
  Paroxysmal Atrial Fibrillation | 1 | 0
  Vasospasm | 1 | 0

4. Secondary Outcome: Assessment of Renovascular Safety as Measured by New Renal Artery Stenosis or Aneurysm at the Site of Ablation
Description: Renovascular safety (new renal artery stenosis or aneurysm) was summarized as a percentage based on the number of subjects at baseline for each group (RDN+AF group= 39, AF group=22).
Time Frame: 6 months and 12 months post procedure
Population: Renovascular safety (new renal artery stenosis or aneurysm) was summarized as a percentage based on the number of subjects at baseline for each group (RDN+AF group= 39, AF group=22).
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Artery Ablation + Cardiac Ablation (RDN+AF) | Cardiac Ablation (AF)
Number analyzed (Participants) | 39 | 22
Participants
  VASC Pseudoaneurysm at 6 months | 1 | 0
  VASC Pseudoaneurysm at 12 months | 2 | 0
  Renal Artery Stenosis at 6 months | 0 | 0
  Renal Artery Stenosis at 12 months | 1 | 0

5. Secondary Outcome: Renal Function Change Based on Estimated Glomerular Filtration Rate (eGFR) (Renal Denervation Group Only) at 6 Months
Time Frame: Baseline and 6 months
Population: eGFR change from baseline was summarized based on subjects with available data at both time points (RDN+AF group = 32)
Measure: Mean (Standard Deviation); unit: mL/min per 1.73m^2
Arm/Group | Renal Artery Ablation + Cardiac Ablation (RDN+AF)
Number analyzed (Participants) | 32
mL/min per 1.73m^2 | 2.2 (11.0)
Statistical Analysis 1: Comparison: Renal Artery Ablation + Cardiac Ablation (RDN+AF); Test type: Superiority; p = 0.2766, Paired Student's t-test

6. Secondary Outcome: Renal Function Change Based on eGFR (Renal Denervation Group Only) at 12 Months
Time Frame: Baseline and 12 months
Population: eGFR change from baseline was summarized based on subjects with available data at both time points (RDN+AF group = 33)
Measure: Mean (Standard Deviation); unit: mL/min per 1.73m^2
Arm/Group | Renal Artery Ablation + Cardiac Ablation (RDN+AF)
Number analyzed (Participants) | 33
mL/min per 1.73m^2 | -0.4 (11.9)
Statistical Analysis 1: Comparison: Renal Artery Ablation + Cardiac Ablation (RDN+AF); Test type: Superiority; p = 0.7663, Wilcoxon signed-rank test

7. Secondary Outcome: Recurrence of Atrial Fibrillation (AF) Based on Electrocardiographic Data up to 2 Years Following the Initial Cardiac Ablation Procedure.
Description: Recurrence of AF was summarized as a percentage based on the number of subjects who underwent the procedure (RDN+AF group= 39, AF group=20)
Time Frame: 3 months, 6 months, 12 months, 24 months
Population: For each group, the outcome measure was analyzed in participants who underwent the procedure (RDN+AF group= 39, AF group=20)
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Artery Ablation + Cardiac Ablation (RDN+AF) | Cardiac Ablation (AF)
Number analyzed (Participants) | 39 | 20
Participants
  Atrial Fibrillation recurrence within 3 months | 4 | 4
  Atrial Fibrillation recurrence within 6 months | 9 | 5
  Atrial Fibrillation recurrence within 12 months | 14 | 8
  Atrial Fibrillation recurrence within 24 months | 19 | 9

8. Secondary Outcome: Percentage of Participants Achieving Office Systolic Blood Pressure < 140 mmHg
Time Frame: 6 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Artery Ablation + Cardiac Ablation (RDN+AF) | Cardiac Ablation (AF)
Number analyzed (Participants) | 35 | 16
Participants | 4 | 1

9. Secondary Outcome: Change in Ambulatory Blood Pressure at 12 Months
Description: Change in Ambulatory Blood Pressure was summarized based on subjects with available data at both time points (RDN+AF group= 22, AF group=14)
Time Frame: Baseline and 12 months post procedure
Population: Change in Ambulatory Blood Pressure was summarized based on subjects with available data at both time points (RDN+AF group= 22, AF group=14)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Artery Ablation + Cardiac Ablation (RDN+AF) | Cardiac Ablation (AF)
Number analyzed (Participants) | 22 | 14
mmHg
  24-Hour Ambulatory Systolic Blood Pressure (ASBP) | -5.9 (15.2) | -3.1 (19.2)
  24-Hour Ambulatory Diastolic Blood Pressure (ADBP) | -5.8 (7.4) | -8.4 (9.4)
Statistical Analysis 1: Comparison: Renal Artery Ablation + Cardiac Ablation (RDN+AF); Change in ASBP at 12 months; Test type: Superiority; p = 0.0849, Paired Student's t-test; Mean Difference (Final Values) = -5.86, 95% CI 2-sided [-12.61 to 0.88], Standard Deviation 15.21
Statistical Analysis 2: Comparison: Renal Artery Ablation + Cardiac Ablation (RDN+AF); Change in ADBP at 12 months; Test type: Superiority; p = 0.0014, Paired Student's t-test; Mean Difference (Final Values) = -5.82, 95% CI 2-sided [-9.12 to -2.52], Standard Deviation 7.45
Statistical Analysis 3: Comparison: Cardiac Ablation (AF); Change in ASBP at 12 months; Test type: Superiority; p = 0.5599, Paired Student's t-test; Mean Difference (Final Values) = -3.07, 95% CI 2-sided [-14.16 to 8.02], Standard Deviation 19.21
Statistical Analysis 4: Comparison: Cardiac Ablation (AF); Change in ADBP at 12 months; Test type: Superiority; p = 0.0052, Paired Student's t-test; Mean Difference (Final Values) = -8.43, 95% CI 2-sided [-13.87 to -2.99], Standard Deviation 9.42

10. Secondary Outcome: Change in Ambulatory Blood Pressure at 24 Months
Description: Change in Ambulatory Blood Pressure was summarized based on subjects with available data at both time points (RDN+AF group= 17, AF group=12)
Time Frame: Baseline and 24 months post procedure
Population: Change in Ambulatory Blood Pressure was summarized based on subjects with available data at both time points (RDN+AF group= 17, AF group=12)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Artery Ablation + Cardiac Ablation (RDN+AF) | Cardiac Ablation (AF)
Number analyzed (Participants) | 17 | 12
mmHg
  24-Hour Ambulatory Systolic Blood Pressure (ASBP) | -5.7 (14.8) | -8.6 (12.4)
  24-Hour Ambulatory Diastolic Blood Pressure (ADBP) | -6.9 (6.1) | -10.3 (8.5)
Statistical Analysis 1: Comparison: Renal Artery Ablation + Cardiac Ablation (RDN+AF); Change in ASBP at 24 months; Test type: Superiority; p = 0.1326, Paired Student's t-test; Mean Difference (Final Values) = -5.71, 95% CI 2-sided [-13.34 to 1.93], Standard Deviation 14.84
Statistical Analysis 2: Comparison: Renal Artery Ablation + Cardiac Ablation (RDN+AF); Change in ADBP at 24 months; Test type: Superiority; p = 0.0002, Paired Student's t-test; Mean Difference (Final Values) = -6.94, 95% CI 2-sided [-10.06 to -3.83], Standard Deviation 6.06
Statistical Analysis 3: Comparison: Cardiac Ablation (AF); Change in ASBP at 24 months; Test type: Superiority; p = 0.0354, Paired Student's t-test; Mean Difference (Final Values) = -8.58, 95% CI 2-sided [-16.47 to -0.70], Standard Deviation 12.41
Statistical Analysis 4: Comparison: Cardiac Ablation (AF); Change in ADBP at 24 months; Test type: Superiority; p = 0.0015, Paired Student's t-test; Mean Difference (Final Values) = -10.33, 95% CI 2-sided [-15.75 to -4.91], Standard Deviation 8.53

11. Secondary Outcome: Change in Office Blood Pressure at 12 Months
Description: Change in Office Blood Pressure was summarized based on subjects with available data at both time points (RDN+AF group= 33, AF group=15)
Time Frame: Baseline and 12 months post procedure
Population: Change in Office Blood Pressure was summarized based on subjects with available data at both time points (RDN+AF group= 33, AF group=15)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Artery Ablation + Cardiac Ablation (RDN+AF) | Cardiac Ablation (AF)
Number analyzed (Participants) | 33 | 15
mmHg
  Change in Office Systolic Blood Pressure (OSBP) | 2.6 (24.4) | 2.0 (30.0)
  Change in Office Diastolic Blood Pressure (ODBP) | -0.4 (11.8) | -5.4 (15.8)
Statistical Analysis 1: Comparison: Renal Artery Ablation + Cardiac Ablation (RDN+AF); Change in OSBP at 12 months; Test type: Superiority; p = 0.5399, Paired Student's t-test; Mean Difference (Final Values) = 2.6, 95% CI 2-sided [-6.0 to 11.3], Standard Deviation 24.4
Statistical Analysis 2: Comparison: Renal Artery Ablation + Cardiac Ablation (RDN+AF); Change in Office Diastolic Blood Pressure (ODBP) at 12 months; Test type: Superiority; p = 0.8489, Paired Student's t-test; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-4.6 to 3.8], Standard Deviation 11.8
Statistical Analysis 3: Comparison: Cardiac Ablation (AF); Test type: Superiority — Change in Office Systolic Blood Pressure (OSBP) at 12 months; p = 0.7999, Paired Student's t-test; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [-14.6 to 18.6], Standard Deviation 30.0
Statistical Analysis 4: Comparison: Cardiac Ablation (AF); Change in ODBP at 12 months; Test type: Superiority; p = 0.2076, Paired Student's t-test; Mean Difference (Final Values) = -5.4, 95% CI 2-sided [-14.2 to 3.4], Standard Deviation 15.8

12. Secondary Outcome: Change in Office Blood Pressure at 24 Months
Description: Change in Office Blood Pressure was summarized based on subjects with available data at both time points (RDN+AF group= 29, AF group=16).
Time Frame: Baseline and 24 months post procedure
Population: Change in Office Blood Pressure was summarized based on subjects with available data at both time points (RDN+AF group= 29, AF group=16).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Artery Ablation + Cardiac Ablation (RDN+AF) | Cardiac Ablation (AF)
Number analyzed (Participants) | 29 | 16
mmHg
  Change in Office Systolic Blood Pressure (OSBP) | 0.6 (22.3) | 7.4 (22.9)
  Change in Office Diastolic Blood Pressure (ODBP) | 0.5 (11.0) | -3.0 (15.5)
Statistical Analysis 1: Comparison: Renal Artery Ablation + Cardiac Ablation (RDN+AF); Change in OSBP at 24 months; Test type: Superiority; p = 0.8820, Paired Student's t-test; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-7.9 to 9.1], Standard Deviation 22.3
Statistical Analysis 2: Comparison: Renal Artery Ablation + Cardiac Ablation (RDN+AF); Change in ODBP at 24 months; Test type: Superiority; p = 0.8019, Paired Student's t-test; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-3.7 to 4.7], Standard Deviation 11.0
Statistical Analysis 3: Comparison: Cardiac Ablation (AF); Change in OSBP at 24 months; Test type: Superiority; p = 0.2177, Paired Student's t-test; Mean Difference (Final Values) = 7.4, 95% CI 2-sided [-4.8 to 19.6], Standard Deviation 22.9
Statistical Analysis 4: Comparison: Cardiac Ablation (AF); Change in ODBP at 24 months; Test type: Superiority; p = 0.4502, Paired Student's t-test; Mean Difference (Final Values) = -3.0, 95% CI 2-sided [-11.2 to 5.2], Standard Deviation 15.5

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Renal Artery Ablation + Cardiac Ablation (RDN+AF) | Cardiac Ablation (AF)
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/22
Serious Adverse Events (participants affected / at risk) | 4/39 | 3/22
Other Adverse Events (participants affected / at risk) | 4/39 | 2/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renal Artery Ablation + Cardiac Ablation (RDN+AF) (N=39) | Cardiac Ablation (AF) (N=22)
Paroxysmal Atrial Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Paroxysmal Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial Tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
VASC Pseudoaneurysm (Vascular disorders) | 1 (1) | 0 (0)
Renal Artery Stenosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renal Artery Ablation + Cardiac Ablation (RDN+AF) (N=39) | Cardiac Ablation (AF) (N=22)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Bleeding (Vascular disorders) | 0 (0) | 1 (1)
Air Embolus (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Vasospasm (Vascular disorders) | 1 (1) | 0 (0)
VASC Pseudoaneurysm (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2014-12-04): https://cdn.clinicaltrials.gov/large-docs/28/NCT01907828/Prot_000.pdf
  • Statistical Analysis Plan (2014-11-05): https://cdn.clinicaltrials.gov/large-docs/28/NCT01907828/SAP_001.pdf